CLINICAL TRIAL: NCT03528603
Title: Acute Assessment of Platelet Reactivity After the Intake of Oleocanthal From Extra Virgin Olive Oil in the Fasted and Fed Condition
Brief Title: Acute Assessment of Platelet Reactivity After the Intake of Oleocanthal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1158686
Record Dates: First submitted 2018-03-27; First posted 2018-05-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2023-05

CONDITIONS: Platelet Aggregation; Nutritional and Metabolic Disease; Cardiovascular Diseases
Keywords: platelet, aggregation, phenolic, olive oil, oleocanthal
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: controlled, randomized, double-blind, with 2 interventions
Who Masked: Participant, Investigator
Masking Description: Extra Virgin Olive Oils will be stored and provided to the study investigators in coded single serving bottles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oleocanthal-Rich Extra Virgin Olive Oil (Experimental): Extra Virgin Olive Oil that is high in the phenolic oleocanthal, but contains similar amounts of total phenolics as the Oleocanthal-Low Extra Virgin Olive Oil
  Interventions: Other: Oleocanthal-Rich Extra Virgin Olive Oil; Other: Oleocanthal-low Extra Virgin Olive Oil
- Oleocanthal-Low Extra Virgin Olive Oil (Placebo Comparator): Extra Virgin Olive Oil that is low in the phenolic oleocanthal, but contains similar amounts of total phenolics as the Oleocanthal-Rich Extra Virgin Olive Oil
  Interventions: Other: Oleocanthal-Rich Extra Virgin Olive Oil; Other: Oleocanthal-low Extra Virgin Olive Oil

INTERVENTIONS:
Other: Oleocanthal-Rich Extra Virgin Olive Oil — Extra Virgin Olive Oil that contains a high level of the phenolic oleocanthal
Other: Oleocanthal-low Extra Virgin Olive Oil — Extra Virgin Olive Oil that contains a low level of the phenolic oleocanthal

SUMMARY:
The investigators have previously observed a reduced level of platelet aggregation 2 hours after healthy male individuals were asked to drink extra virgin olive oil (EVOO) that provided a higher level of one specific phenolic known as oleocanthal. This study will help the investigators further determine the effects of oleocanthal-rich EVOO intake on platelet function at 2, 4 and 6 hours after intake with food compared to platelet function in the morning after an overnight fast.

DETAILED DESCRIPTION:
Fifty adult male volunteers will be asked to participate in one of two study trials that will be randomized double-blind controlled crossover trials with 2 study visits. The participants will arrive to the facility after an overnight fast, and will be asked to consume their assigned EVOO either without (trial 1) or with (trial 2) a standardized low-phenolic food (such as rice, pasta or mashed potatoes) with 40 mL of one of 2 EVOOs that are matched for their total phenolic content, but with one oil containing oleocanthal, and one with very low levels of oleocanthal. At zero, two, 4 and 6 hours after EVOO intake a blood sample will be collected for the assessment of collagen- ADP-, and AA-induced platelet aggregation, as well as an untargeted metabolomics profile.

As an assessment of phenotypic stability, a subset of individuals (n=5 per trial) that have exhibit either low or high platelet responses, will be asked to repeat the above study.

ELIGIBILITY:
Inclusion Criteria:

* Trials 1 and 2: Male; Trial 3: Male and Female
* 20-45 years old
* For females, a regular 25-30-day menstrual cycle
* Subject is willing and able to comply with the study protocols
* Subject is willing to drink 40 mL (approximately 2 tablespoons) of olive oil
* BMI 18.5 - 30 kg/m2
* Weight ≥ 110 pounds

Exclusion Criteria:

* Adults who are not able to consent
* BMI ≥ 31 kg/m2
* Under current medical supervision
* 1 ug/ml and 3 ug/ml collagen screening maximal platelet aggregatory response of < 65%.
* Platelet number or mean platelet values that are outside of the normal reference range as indicated on a complete blood cell count report from the UCD Med Center
* Current diagnosis of anemia; or a screening hemoglobin and hematocrit that is less than the normal reference range.
* Self-reported daily use of drugs that are known to affect platelet function, such as aspirin, Excedrin, and NSAIDS
* Females using hormonal contraception
* Ibuprofen intolerance or allergy
* Those with a bleeding disorder
* Non-English speaking
* Allergy to olives or olive oil
* Vegetarian, Vegan, food faddists, individuals using non-traditional diets, or on a weight loss diet.
* A history of cardiovascular disease, stroke, cancer, renal, hepatic, or thyroid disease, GI tract disorders, previous GI surgery
* Currently taking prescription drugs or supplements
* Indications of substance or alcohol abuse within the last 3 years
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements for six weeks prior to study enrollment.
* Not willing to refrain from olive oil consumption for 4 weeks prior to study enrollment, and throughout study enrollment
* Self-reported malabsorption (e.g. difficulty digesting or absorbing nutrients from food, potentially leading to bloating, cramping or gas)
* Current enrollee in a clinical research study.
* Individuals with blood clotting or platelet defect disorders

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Influence of Oleocanthal-rich EVOO intake on Collagen-induced platelet aggregometry | baseline, 2, 4 and 6 hours
  Optical platelet aggregometry will be used to measure platelet aggregation. The percent maximal platelet aggregation will be measured. A reduction in maximal aggregation 2, 4 or 6 hours post EVOO intake compared to baseline will represent a reduction in platelet aggregation.

SECONDARY OUTCOMES:
Influence of Oleocanthal-rich EVOO intake on Adenosine Diphosphate-induced platelet aggregometry | baseline, 2, 4 and 6 hours
  Optical platelet aggregometry will be used to measure platelet aggregation. The percent maximal platelet aggregation will be measured. A reduction in maximal aggregation 2, 4 or 6 hours post EVOO intake compared to baseline will represent a reduction in platelet aggregation.
Influence of Oleocanthal-rich EVOO intake on Arachidonic Acid-induced platelet aggregometry | baseline, 2, 4 and 6 hours
  Optical platelet aggregometry will be used to measure platelet aggregation. The percent maximal platelet aggregation will be measured. A reduction in maximal aggregation 2, 4 or 6 hours post EVOO intake compared to baseline will represent a reduction in platelet aggregation.
Influence of Oleocanthal-rich EVOO intake on Platelet-derived oxylipins | baseline, 2, 4 and 6 hours
  Oxylipin profile will be conducted from the activated platelet supernatant ultra high-performance liquid chromatography-mass spectrometry (HPLC) is used to measure levels of oxylipin. HPLC area under the peak will be measured.
Influence of Oleocanthal-rich EVOO intake on Metabolomics | baseline, 2, 4 and 6 hours
  Untargeted metabolomics will be performed to assess the relationship between platelet response and the presence of circulating plasma metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/study-of-the-effects-of-extra-virgin-olive-oil-polyphenols-on-cardiovascular-health-162282/